CLINICAL TRIAL: NCT03830138
Title: Oxidized LDL, Oxidized LDL Receptor 1 (OLR1) Gene Polymorphism With Oxygen Therapy in Acute Myocardial Infarction.
Brief Title: Oxidized LDL With Oxygen Therapy in Acute Coronary Syndrome.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Acute coronary syndrome
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Oxidized-LDL; OLR1 gene; Single nucleotide polymorphism; Oxygen therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute coronary syndrome patients:: One hundred patients with acute coronary syndrome.
  Interventions: Genetic: Oxidized-LDL gene polymorphism
- Controls:: Fifty healthy control
  Interventions: Genetic: Oxidized-LDL gene polymorphism

INTERVENTIONS:
Genetic: Oxidized-LDL gene polymorphism — Oxidized-LDL gene polymorphism will be measured by RFLP. In addition, Oxidized-LDL will be measured in the plasma by ELISA

SUMMARY:
Coronary artery disease (CAD) is increasing rapidly in Egyptian people and manifesting a younger age. Higher plasma low-density lipoprotein cholesterol (LDL-C), is a major predictor for the development of CAD. However, whether oxidized-LDL (ox-LDL) can be used as a risk factor for myocardial infarction (MI) has not been fully investigated. Therefore, the aim of the present study was to examine the role of ox-LDL as a risk factor for the presence and clinical outcomes in patients with MI.

DETAILED DESCRIPTION:
Cardiovascular disease, which is multifactorial and caused by complex interactions of genetic and environmental factors, represents the main cause of death all over the world. Traditional risk factors for coronary atherosclerosis include age, smoking, male gender, hypertension and diabetes. Newly defined risk factors such as hyper-homocysteine, elevated plasma levels of OxLDL and oxidative stress are also emerging.

Lectin-like oxidized low-density lipoprotein receptor-1 (LOX-1) is the major receptor of oxidized low-density lipoproteins which regulates the growth of a variety of cells and is important in inflammation, atherosclerosis, oxidative stress, and tissue remodeling. LOX-1 is expressed in various cells, including endothelial cells, macrophages, and chondrocytes, and its expression is enhanced by proinflammatory cytokines. The LOX1 gene, also known as OLR1, is located on the chromosome 12p13.1-p12.3. The LOX1 protein is synthesized as a 40-kDa precursor protein and is composed of four domains: an extracellular lectin-like domain at the C-terminal, a connecting neck domain, a transmembrane domain, and an N-terminal cytoplasmic domain. Three single nucleotide polymorphism (SNPs), namely, intron 4 (G→A), intron 5(T→G), and 3' UTR (T→C) in the LOX1 gene, have been previously reported. These polymorphisms have also been associated with CAD.

Oxygen is a lifesaving drug. Giving oxygen to a patient with an impending clinical emergency has become knee-jerk reflex reaction of the clinician. Patient with AMI has compromised myocardial perfusion and event arises due to myocardial hypoxia. It appears quite logical and biologically plausible to give oxygen in such situations to improve the oxygenation of the ischemic myocardial tissue and decrease ischemic pain. On the other side, oxygen may be harmful with a mechanism such as the paradoxical effect of oxygen in decreasing coronary artery blood flow and increasing coronary vascular resistance due to increased oxygen free radicals. The investigators aimed to examine the association of the OLR1 gene with AMI or CAD in a novel, well-phenotyped, and homogenous, population and its correlation with oxygen therapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included irrespective of concomitant risk factors for atherosclerosis such as smoking, arterial hypertension and diabetes mellitus.
* Participants were both sexes.

Exclusion Criteria:

* Congenital heart disease.
* Dilated, hypertrophic or restrictive cardiomyopathy.
* acute and chronic liver disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acute coronary syndrome patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
The mean difference of oxidized-LDL gene polymorphism between patients and controls | Baseline
  The mean difference of oxidized-LDL gene polymorphism will be assessed by RFLP. The change of single nucleotide polymorphism of oxidized-LDL from healthy controls at baseline

REFERENCES:
- [Background] Ehara S, Ueda M, Naruko T, Haze K, Itoh A, Otsuka M, Komatsu R, Matsuo T, Itabe H, Takano T, Tsukamoto Y, Yoshiyama M, Takeuchi K, Yoshikawa J, Becker AE. Elevated levels of oxidized low density lipoprotein show a positive relationship with the severity of acute coronary syndromes. Circulation. 2001 Apr 17;103(15):1955-60. doi: 10.1161/01.cir.103.15.1955. PMID 11306523
- [Background] Trabetti E, Biscuola M, Cavallari U, Malerba G, Girelli D, Olivieri O, Martinelli N, Corrocher R, Pignatti PF. On the association of the oxidised LDL receptor 1 (OLR1) gene in patients with acute myocardial infarction or coronary artery disease. Eur J Hum Genet. 2006 Jan;14(1):127-30. doi: 10.1038/sj.ejhg.5201513. PMID 16251892
- [Background] Zhao X, Zhang HW, Xu RX, Guo YL, Zhu CG, Wu NQ, Gao Y, Li JJ. Oxidized-LDL is a useful marker for predicting the very early coronary artery disease and cardiovascular outcomes. Per Med. 2018 Nov;15(6):521-529. doi: 10.2217/pme-2018-0046. Epub 2018 Oct 26. PMID 30362886
- [Background] Raut MS, Maheshwari A. Oxygen supplementation in acute myocardial infarction: To be or not to be? Ann Card Anaesth. 2016 Apr-Jun;19(2):342-4. doi: 10.4103/0971-9784.179594. No abstract available. PMID 27052081